CLINICAL TRIAL: NCT00003070
Title: Afterload Reduction Therapy for Late Anthracycline Cardiotoxicity: A Pediatric Oncology Group Cancer Control Study
Brief Title: Enalapril in Treating Heart Damage Patients Who Received Anthracycline Chemotherapy for Childhood Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: P9480; POG-9480 (Other: Pediatric Oncology Group); NCI-P97-0086 (Other: NCI Trial Identifier); CDR0000065745 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Toxicity; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; cardiac toxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Stratum 1 < 350/mg/m2 anthracycline dose (Experimental): < 4 years of age at diagnosis < 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 2 < 350mg/m2 anthracycline dose (Experimental): < 4 years of age at diagnosis >= 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 3 < 350mg/m2 anthracycline dose (Experimental): >= 4 years of age at diagnosis < 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 4 < 350mg/m2 anthracycline dose (Experimental): >= 4 years of age at diagnosis >= 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 5 >= 350mg/m2 anthracycline dose (Experimental): < 4 years of age at diagnosis < 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 6 >=350mg/m2 anthracycline dose (Experimental): < 4 years of age at diagnosis < 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 7 >= 350mg/m2 anthracycline dose (Experimental): >= 4 years of age at diagnosis < 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment
- Stratum 8 >= 350mg/m2 anthracycline dose (Experimental): >= 4 years of age at diagnosis >= 4 years since cessation of anthracycline treatment
  Interventions: Drug: enalapril maleate; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: enalapril maleate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as enalapril, may protect normal cells from the toxic effects of chemotherapy. It is not known whether enalapril is more effective than a placebo in treating heart damage in patients who received anthracycline chemotherapy for childhood cancer.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of enalapril with a placebo in treating heart damage in patients who received anthracycline chemotherapy for childhood cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether enalapril treatment results in a reduction in body surface area-adjusted left ventricular mass in anthracycline-treated survivors of childhood cancer. II. Determine whether improvement in ventricular function achieved by enalapril is sustained and alters the course of late cardiotoxicity. III. Determine the impact of enalapril therapy on quality of life.

OUTLINE: This is a double blind, placebo controlled, randomized study. Patients are stratified based on the cumulative anthracycline dose, age at cancer diagnosis, and the duration of time since cessation of anthracycline therapy. Patients are administered enalapril or placebo by mouth bid. Patients undergo a series of cardiac tests after administration of drug. Follow-up occurs at 2, 6, and 12 months and every year thereafter.

PROJECTED ACCRUAL: 75 patients in each treatment arm will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed childhood malignancy that had prior anthracycline therapy Echocardiographic evidence of reduced fractional shortening, reduced contractility, or increased afterload, or any combination At least 6 months oncologic disease free

PATIENT CHARACTERISTICS: Age: At least 8 at study entry and less than 22 at diagnosis Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: No history of renal disease No known renal artery stenosis Cardiovascular: No congenital cardiovascular malformations No active congestive heart failure not attributable to sepsis or renal failure No medication for heart condition No history of symptomatic arrhythmia antedating anthracycline therapy No constrictive pericarditis No uncontrolled hypertension Pulmonary: No primary valvular or outflow tract obstruction Other: Not pregnant or lactating Must use adequate contraception No reaction or intolerance to ACE inhibitors

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 1 year since prior cumulative anthracycline therapy of at least 200 mg/m2 No prior amsacrine therapy Endocrine therapy: Not specified Radiotherapy: No prior mediastinal, spinal, or total body irradiation that included the heart Surgery: Not specified Other: No concurrent angiotensin converting enzyme (ACE)inhibitor treatment No concurrent treatment with other investigational drug No oncologic therapy within past 6 months

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2000-09; Primary Completion 2003-07 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Cardiac functional status and quality of life | baseline, two and five years
  Cardiac functional status (depressed fractional shortening) and quality-of-life, will be assessed at baseline, two and five years into the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lipshultz, MD, Study Chair — James P. Wilmot Cancer Center
Locations (61):
- United States (55):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Children's Hospital, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- Swiss Pediatric Oncology Group Bern, Bern, Switzerland

REFERENCES:
- [Background] Krischer JP, Epstein S, Cuthbertson DD, Goorin AM, Epstein ML, Lipshultz SE. Clinical cardiotoxicity following anthracycline treatment for childhood cancer: the Pediatric Oncology Group experience. J Clin Oncol. 1997 Apr;15(4):1544-52. doi: 10.1200/JCO.1997.15.4.1544. PMID 9193351